CLINICAL TRIAL: NCT01651377
Title: Pramipexole as a Treatment for Cocaine Dependence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Thomas Newton, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: H-28454; 5P50DA018197 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2012-02-20; First posted 2012-07-27 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Cocaine Addiction; Cocaine Abuse; Cocaine Dependence; Substance Abuse
Keywords: Pramipexole; Mirapex; Cocaine
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Pramipexole; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Pramipexole (Active Comparator)
  Interventions: Drug: Pramipexole

INTERVENTIONS:
Drug: Pramipexole — Participants will receive pramipexole ER 0.375, .075, 1.5, 2.25, and 3mg/d in an ascending-dose pattern.
  Other Names: Mirapex
  Arms: Pramipexole
Drug: Placebo — Participants will receive matching placebo pills. The placebo group is included to maintain the blind, rather than as a comparison group.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The purposes of this study are as follows: 1. To assess the cardiovascular and subjective effects of cocaine during treatment with pramipexole and placebo. 2. To assess the reinforcing effects of cocaine, measured using choice procedures, during treatment with pramipexole and placebo.

DETAILED DESCRIPTION:
In this protocol we propose to assess the impact of treatment with higher doses of the potent D2/3 agonist pramipexole, using the extended release preparation that has been shown to produce continuous DA receptor stimulation. Pramipexole is a non-ergot DA 3 receptor-preferring agonist. In contrast to pergolide, bromocriptine and cabergoline, it does not stimulate 5-HT2B receptors and therefore does not cause cardiac valvulopathy. It can therefore be safely used chronically at higher doses, whereas pergolide has been withdrawn from the market for causing cardiac valvulopathy.

ELIGIBILITY:
Inclusion Criteria:

* Be English-speaking volunteers who are not seeking treatment at the time of the study. We require proficiency in English to ensure good communication with staff.
* Be aged between 18 and 55 years.
* Meet DSM-IV TR criteria for cocaine dependence.
* Have a self-reported history of using cocaine by the IV or smoked route.
* Have vital signs as follows: supine blood pressure > 100/65 mm Hg, a seated blood pressure of > 90/60 mm Hg, and an orthostatic change < 20 mm Hg systolic or <10 mm Hg diastolic on standing. To ensure that subjects will not be at risk from cocaine, the resting pulse must be < 90 bpm and the blood pressure must be < 150 mmHg systolic and < 90 mmHg diastolic.
* Have hematology and chemistry laboratory tests that are within reference limits (±10%), with the following exceptions: (a) total bilirubin must be < 2x upper limit of normal and ALT, AST, and alkaline phosphatase <3× the upper limit of normal and (b) kidney function tests (creatinine and BUN) within normal limits.
* Have a baseline ECG that demonstrates clinically normal sinus rhythm, clinically normal conduction, and no clinically significant arrhythmias.
* Have a medical history and brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the admitting physician and the principal investigator.

Exclusion Criteria:

* Have any history or evidence suggestive of seizure disorder or brain injury.
* Have any previous medically adverse reaction to cocaine, including loss of consciousness, chest pain, or epileptic seizure.
* Have neurological or psychiatric disorders, such as: psychosis, bipolar illness or major depression as assessed by SCID; organic brain disease or dementia assessed by clinical interview; history of any psychiatric disorder that would require ongoing treatment or that would make study compliance difficult; and history of suicide attempts within the past year and/or current suicidal ideation/plan.
* Have evidence of clinically significant heart disease or hypertension, as determined by the PI.
* Have a family history in first-degree relatives of early cardiovascular morbidity or mortality, as determined by the PI.
* Have evidence of untreated or unstable medical illness including neuroendocrine, autoimmune, renal, hepatic, or active infectious disease.
* Have HIV and are currently symptomatic or are taking antiretroviral medication.
* Be pregnant or nursing. Females must provide negative pregnancy urine tests upon hospital admission and at the end of study participation. Females must either be unable to conceive (i.e., surgically sterilized, sterile, or postmenopausal) or be using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device, or condoms with spermicide).
* Have asthma or currently use theophylline or other sympathomimetics.
* Have any other illness, condition, or use of psychotropic medications, which in the opinion of the PI and/or the admitting physician would preclude safe and/or successful completion of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The effects of pramipexole and cocaine on cardiovascular measures | 16 days
  Before and after each cocaine infusion, physiologic responses will be closely monitored using repeated HR, BP, and ECG readings. To evaluate safety, a DSMB will meet annually and following any serious AE to examine data as well as any new published information on pramipexole relevant to the project. The number of AEs (including arrhythmias and ECG changes), changes in BP and HR, and changes in mood and psychiatric symptoms (using the BSI, BDI, POMS, and BPRS) will also be assessed throughout the study.

SECONDARY OUTCOMES:
The effects of pramipexole and cocaine on subjective measures | 16 days
  The ability of pramipexole, as compared to placebo, to reduce cocaine-induced craving and to reduce reinforcing effects produced by cocaine will be measured by: 1. VAS, Adjective Scales, and MCQ; 2. Choices for cocaine vs. money in the self-administration assay.

CONTACTS AND LOCATIONS:
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States

REFERENCES:
- [Derived] Newton TF, Haile CN, Mahoney JJ 3rd, Shah R, Verrico CD, De La Garza R 2nd, Kosten TR. Dopamine D3 receptor-preferring agonist enhances the subjective effects of cocaine in humans. Psychiatry Res. 2015 Nov 30;230(1):44-9. doi: 10.1016/j.psychres.2015.07.073. Epub 2015 Jul 29. PMID 26239766